CLINICAL TRIAL: NCT05308953
Title: A Randomized, Triple-Blind, Placebo-Controlled Phase I Study of Single and Multiple Ascending Doses of NVG-291 in Healthy Subjects
Brief Title: A Phase I Safety Study of NVG-291 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NervGen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: NVG-291-101
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NVG-291 SAD (Experimental): Doses will begin at the lowest dose level in Cohort 1, increasing in dose with each subsequent cohort to the highest dose level in Cohort 6 or until a maximum tolerated dose (MTD) is reached.
  Interventions: Drug: NVG-291; Other: Placebo
- NVG-291 MAD (Experimental): Participants will receive 1 dose daily for for 14 consecutive days. The maximum starting dose for MAD will be 2 dose levels lower than the maximum dose achieved during SAD. There will be a maximum of 3 dosing cohorts in Part 2. The maximum daily dose in Part 2 will not exceed the maximum daily dose tolerated in Part 1.
  Interventions: Drug: NVG-291; Other: Placebo
- NVG-291 MAD - Males and Premenopausal Females (Experimental): Participants will receive 1 dose daily for for 14 consecutive days. The dose maximum daily dose in Part 3 will not exceed the maximum daily dose tolerated in either Part 1 or 2.
  Interventions: Drug: NVG-291; Other: Placebo

INTERVENTIONS:
Drug: NVG-291 — NVG-291 is a drug injected under the skin (subcutaneous).
Other: Placebo — Salt water is being used as a placebo and will be injected under the skin (subcutaneous).

SUMMARY:
This is a randomized, triple-blind (subjects, Investigators, and Sponsor blinded), placebo-controlled Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) study to evaluate the safety and tolerability of NVG-291 administered by subcutaneous injection daily in healthy female participants. The trial is split into three parts, starting with Part 1 (SAD), then Part 2 (MAD - post-menopausal Females), and finally Part 3 (MAD - males and premenopausal females). In Part 1 (SAD), participants receive 1 dose on 1 day only and in Parts 2 and 3, participants receive 1 dose every day for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between 18 and 65 years old.
2. BMI between 18 and 33 kg/m2, inclusive, and a total body weight > 50 kg.
3. All laboratory values must be within normal limits or any abnormalities deemed not clinically significant.
4. All subjects must be willing to abstain from sexual intercourse or to use adequate contraception during the study and for an additional 120 days after the follow-up visit.
5. Subjects must not donate ova or sperm during the study and for an additional 120 days after the follow-up visit
6. Subjects must be willing and able to comply with scheduled visits, all sample collections, and other trial procedures.
7. Subjects must provide written informed consent.

Exclusion Criteria:

1. For premenopausal female subjects: Irregular menstrual cycles; Amenorrhea; or Abnormal vaginal bleeding
2. A history (within the past year) or presence of a clinically significant infectious disease or hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, neurologic, or psychiatric abnormality.
3. Blood pressure > 160/95 at screening or on Day -1.
4. Any active or uncontrolled infections or other medical condition or circumstance that could interfere with the subject's participation in the study.
5. History of allergic reaction to mannitol.
6. Presence of a tattoo, piercing, scar, or other dermatologic abnormality at the injection site (abdomen), that might interfere with the ability to assess injection site reactions
7. a significant history of atopic dermatitis as an adult, or history of severe allergic reaction to injections.
8. INR > 1.4 or PTT > 50 or platelets <50x10^3/µL at screening or on Day -1.
9. History of regular alcohol consumption exceeding 10 units/week (1 unit = 83 mL of 12% wine) within 6 months of screening.
10. Test positive for use of drugs or alcohol at screening.
11. Positive hepatitis B, hepatitis C, or HIV test at screening.
12. Blood or plasma donation within 1 week prior to Day -1.
13. Receipt of an investigational drug within 30 days or five half-lives of the drug (whichever is longer) prior to Day -1.
14. Prior participation in this trial.
15. Female subjects who are breastfeeding or who have a positive pregnancy test at screening or Day -1.
16. History of any condition that might impair the subject's ability to understand or to comply with the requirements of the study or to provide informed consent.
17. Receipt of a COVID-19 vaccination within 3 weeks prior to Day -1
18. Subject is at risk of self-harm or harm to others as evidenced by past suicidal behavior or endorsing items 4 or 5 on the Columbia-Suicide Severity Rating Scale at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-06-04 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Assessed through 7 days following the last dose of study drug
  number and frequency of adverse events

SECONDARY OUTCOMES:
Pharmacokinetic analysis (plasma) | Assessed on Day 1 (SAD and MAD) and Day 14 (MAD only)
  measure of concentration of drug in blood plasma
Immunogenicity analysis | Assessed on Day 1 (SAD and MAD), Day 8 (SAD and MAD) and Day 21 (MAD only)
  number of participants with confirmed and titer results for the presence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Miko, MD, Study Director — CMO
Locations (1):
- Nucleus Networks, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No